CLINICAL TRIAL: NCT04924894
Title: Determinants of Obtaining COVID-19 Vaccination Among Health Care Workers Accessible to Free COVID-19 Vaccination: a Cross Sectional Study
Brief Title: Determinants of Obtaining Covid Vaccination Among Health Care Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maiada K. Hashem, Lecturer, Assiut University
Other Study IDs: Attitude towards COVID vaccine
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Vaccination
Keywords: COVID-19, Vaccine, acceptance, attitude
MeSH Terms: conditions — COVID-19; Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Despite the global preventive efforts (physical distancing, face, mask, travel constraints, and quarantine) to contain the infection, COVID-19 is continuing with its devastating consequences on health, life, and economics. The world's hopes are attached to a successful preventive measure that is the vaccination which has proved its capability to stop infections and save lives over the years. World Health Organization (WHO) declared vaccination hesitancy as one of the top 10 obstacles for global health. Multicentric study involved Arab countries measure hesitancy of HCWs toward vaccine, it reported the highest rates of hesitancy were among participants from the western regions of the Arab world (Egypt, Morocco, Tunisia, and Algeria). This study aims to evaluate the attitude and the determinants of this attitude of HCWs towards receiving or refusing to have their first dose of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* All staff how are working in AUH and offered to receive the first dose of AstraZeneca & Sino pharm vaccine.

Exclusion Criteria:

* Those who are not eligible to receive the vaccine
* Those who are not freely offered to receive the vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthcare workers in Assiut university hospitals how are eligible for COVID-19 vaccination and the vaccine is freely offered to them
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
The rate of acceptance among HCWs who offered COVID-19 vaccine | baseline
  to evaluate the rate of acceptance or refusal of receiving COVID-19 vaccines among health care workers

SECONDARY OUTCOMES:
1. Reasons for acceptance 2. Reasons for refusal 1. Reasons for acceptance 2. Reasons for refusal the response for COVID-19 vaccination acceptance or refusal | baseline
  to understand the causes of vaccination acceptance or refusal among HCWs

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qunaibi E, Basheti I, Soudy M, Sultan I. Hesitancy of Arab Healthcare Workers towards COVID-19 Vaccination: A Large-Scale Multinational Study. Vaccines (Basel). 2021 May 2;9(5):446. doi: 10.3390/vaccines9050446. PMID 34063313
- [Background] Pogue K, Jensen JL, Stancil CK, Ferguson DG, Hughes SJ, Mello EJ, Burgess R, Berges BK, Quaye A, Poole BD. Influences on Attitudes Regarding Potential COVID-19 Vaccination in the United States. Vaccines (Basel). 2020 Oct 3;8(4):582. doi: 10.3390/vaccines8040582. PMID 33022917